CLINICAL TRIAL: NCT04332939
Title: Activating Motor System to Relieve Pain in Elderly: What is the Role of Physical Exercise and Transcranial Stimulation
Brief Title: Motor System Activation With Transcranial Direct Current Stimulation and Physical Exercise to Reduce Pain in Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Guillaume Léonard, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-3273
Record Dates: First submitted 2020-01-23; First posted 2020-04-03 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pain
Keywords: transcranial direct current stimulation; physical exercise; corticospinal projections
MeSH Terms: conditions — Chronic Pain; Motor Activity | interventions — Transcranial Direct Current Stimulation; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + real tDCS (Experimental): Intervention will last 8 weeks where participants will be trained at a rate of 3 workouts per week.
  For the first week, participants will receive 5 daily sessions of anodal tDCS (2 mA, 20 min).
  Interventions: Other: transcranial direct current stimulation; Other: Physical exercise
- Exercise + Sham tDCS (Sham Comparator): Intervention will last 8 weeks where participants will be trained at a rate of 3 workouts per week.
  For the first week, participants will receive 5 daily sessions of sham tDCS.
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: transcranial direct current stimulation — real tDCS sessions
  Arms: Exercise + real tDCS
Other: Physical exercise — Aerobic exercise and physical training combined with sham tDCS

SUMMARY:
Physical exercises are known to reduce chronic pain in elderly individuals by activating the motor system. However, it seems that exercises are not effective for everyone. The investigators believe that elderly individuals with altered corticospinal tract will be those in whom the exercise alone are not sufficient to relieve pain. For those patients, adding an exogenous stimulation of the motor system such as transcranial direct current stimulation (tDCS) would facilitate the corticospinal tract, and consequently, would help exercises to relieve chronic pain. The investigators hypothesize that combining tDCS with the exercises will be more effective than exercises alone, but only in individuals who initially show low corticospinal projections.

DETAILED DESCRIPTION:
Prevalence and intensity of chronic pain increases substantially with age. According to several studies, physical exercises are effective to reduce chronic pain in elderly. However, it seems that exercises are not effective for everyone. One of the hypotheses raised is that the people in whom the exercises have no effect would be those with an alteration of the corticospinal tract. Transcranial direct current stimulation (tDCS) is a non-invasive neurostimulation technique known to facilitate the corticospinal tract when applied over the motor cortex.

Elderly suffering from chronic pain will be recruited in this double-blind, parallel-group, randomised control trial. Participants will be randomized to receive exercises combined to real tDCS (5 daily sessions, 2 mA, 20 minutes) or to sham tDCS. Intervention will last 8 weeks at a rate of 3 workouts per week.

ELIGIBILITY:
Inclusion Criteria:

* To have musculoskeletal chronic pain
* Not to change medication and life habits during the study

Exclusion Criteria:

* People physically active before the study (more then 150 min of moderate to vigorous exercise par week)
* To have an uncontrolled cardiovascular disease
* To have orthopedic limitation or contraindication to physical exercise
* To have contraindication to tDCS
* To have contraindication to TMS
* To have contraindication to MRI

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain intensity | Before intervention (T1), First week of intervention (T2), Week 4 (T3), Week 8 (T4), Follow-up 1 week after intervention (T5), Follow-up 1 month after intervention (T6)
  Pain intensity will be assessed with a pain logbook containing a numerical rating scale from 0 to 10

SECONDARY OUTCOMES:
Corticospinal excitability (TMS) | Before intervention, Follow-up 1 week after, Follow-up 1 month after
  Corticospinal tract excitability will be assessed with transcranial magnetic stimulation (TMS)
Corticospinal excitability (dMRI) | Before intervention, Follow-up 1 week after, Follow-up 1 month after
  Corticospinal tract excitability will be assessed diffusion magnetic resonance imaging
Functional connectivity | Before intervention, Follow-up 1 week after intervention, Follow-up 1 month after intervention
  Functional connectivity will be assessed with functional magnetic resonance imaging
McGill pain questionnaire | Before intervention, Follow-up 1 week after intervention, Follow-up 1 month after intervention
  McGill pain questionnaire will be used to assess pain in its globality. Score from 0 to 72, higher score means worse outcome.
Brief pain inventory | Before intervention, Follow-up 1 week after intervention, Follow-up 1 month after intervention
  Brief pain inventory will be used to assess pain in its globality. Score from 0 to 70, higher score means worse outcome
Beck depression inventory | Before intervention, Follow-up 1 week after intervention, Follow-up 1 month after intervention
  Beck depression inventory will be used to assess pain in its globality. Score from 0 to 39, higher score means worse outcome
Beck anxiety inventory | Before intervention, Follow-up 1 week after intervention, Follow-up 1 month after intervention
  Beck anxiety inventory will be used to assess pain in its globality. Score from 0 to 63, higher score means worse outcome
Margolis pain drawing and scoring system | Before intervention, Follow-up 1 week after intervention, Follow-up 1 month after intervention
  Margolis pain drawing and scoring system will be used to assess pain in its globality. Score from 0 to 45, higher score means worse outcome
Patient global impression of change questionnaire | Before intervention, Follow-up 1 week after intervention, Follow-up 1 month after intervention
  patient global impression of change questionnaire will be used to assess pain in its globality. Score from 0 to 18 and a percentage from 0 to 100. Higher scores mean better outcome
Tampa questionnaire | Before intervention, Follow-up 1 week after intervention, Follow-up 1 month after intervention
  Tampa questionnaire will be used to assess pain in its globality. Score from 0 to 68, higher score means worse outcome
Pain catastrophizing scale | Before intervention, Follow-up 1 week after intervention, Follow-up 1 month after intervention
  Pain catastrophizing scale will be used to assess pain in its globality. Score from 0 to 52, higher score means worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Léonard, pht, PhD., Principal Investigator — Université de Sherbrooke
Locations (2):
- Canada (2):
  - Research Centre on Aging, Sherbrooke, Quebec
  - Grace Village, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No